CLINICAL TRIAL: NCT05169229
Title: Antibiotic Impregnated Bone Graft to Reduce Infection in Hip Replacement. The ABOGRAFT Trial
Brief Title: Antibiotic Impregnated Bone Graft to Reduce Infection in Hip Replacement.
Acronym: ABOGRAFT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Region Östergötland (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Jörg Schilcher, Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABOGRAFT-01; 2021-001708-14 (EudraCT Number)
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Arthroplasty, Replacement, Hip; Osteoarthritis, Hip; Antibiotic Resistant Infection; Prosthetic Joint Infection
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Vancomycin; Tobramycin; Therapeutics; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A pragmatic, phase II, randomized, double-blind, placebo-controlled, multicenter drug trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Combination of vancomycin and tobramycin mixed with allograft and locally administered during revision surgery after total hip arthroplasty.
  Interventions: Drug: Vancomycin + Tobramycin
- Placebo (Placebo Comparator): Saline locally added to allograft and locally administered during revision surgery after total hip arthroplasty.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Vancomycin + Tobramycin — 1 g vancomycin (powder) diluted in 8 ml tobramycin (40 -80mg/ml). Added to the prepared allograft before the allograft is used during the revision surgery.
  Other Names: Treatment
  Arms: Treatment arm
Drug: Saline — As a placebo added to the allograft.
  Other Names: Control
  Arms: Placebo

SUMMARY:
Total hip replacement is the most successful treatment modern healthcare can offer patients to regain quality of life. Periprosthetic joint infection (PJI) is the most common and devastating complication after total hip replacement (THR). Between 0.5 to 2% of primary THR (first time hip replacement), and 8-10% of revision THR (replacement of a hip prosthesis) will become infected.1 The introduction of local antibiotics blended into bone cement has led to a reduction in postoperative infection in primary THR by half.2 Unfortunately, cement can't always be used in relevant quantities.

The number of primary and revision surgeries of the hip is projected to increase dramatically. Therefore, the need for a feasible infection prophylaxis that is applicable for complex primary and revision THR in addition to antibiotics loaded cement is urgent.

Impacted morselized bone allograft is often used in (revision) THR to fill bone defects. Morselized allograft has been used as a carrier for local antibiotic treatment in multiple pilot studies and appears to be an attractive and effective treatment option, both for already infected joints and as a prophylactic measure in high-risk patients (e.g. THR revision surgeries). Nonetheless, a pivotal trial to support its use in THR is lacking. The aim of this pragmatic randomized controlled double blinded drug trial is to investigate whether antibiotic impregnated bone graft (AIBG) decreases the risk of infection after hip arthroplasty compared to controls treated with placebo impregnated bone graft. Patients scheduled for elective THR will be randomized to receive AIBG or a placebo impregnated bone graft. The primary outcome variable will be the number of re-operations due to infections and PJI diagnoses 2 years postoperative.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Hip arthroplasty requiring bone graft
3. Willing to provide informed consent.
4. For women of childbearing potential; a negative pregnancy test prior to reoperation.

Exclusion Criteria:

1. Ongoing prosthetic joint infection
2. Known allergies and contraindications for the use of vancomycin or tobramycin
3. Mental inability, reluctance, or language difficulties that according to investigator judgement, result in difficulty understanding the meaning of study participation
4. Expected difficulties to complete 2-year follow-up
5. Females of child bearing potential not using contraception
6. Pregnant females
7. Nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Reoperation due to infection or diagnosed PJI with bacteria that are sensitive to either vancomycin or tobramycin, in the same hip joint, within two years after hip arthroplasty. | 2 years after finalizing data collection.
  Reoperation due to infection or diagnosed PJI 2 years of revision surgery.

SECONDARY OUTCOMES:
Time and cause for reoperation for any reason within 2 and 5 years | 2 and 5 years after finalizing data collection.
  Time and cause for reoperation for any reason within 2 and 5 years
Time and cause for implant revision due to any reason within 2 and 5 years | 2 and 5 years after finalizing data collection.
  Time and cause for implant revision due to any reason within 2 and 5 years
Type of microbe and antibiotic resistance pattern for cases complicated with postoperative infection | 2 and 5 years after finalizing data collection.
  Type of microbe and antibiotic resistance pattern for cases complicated with postoperative infection

OTHER OUTCOMES:
Differences between the two experimental groups regarding the frequencies of adverse events | 2 and 5 years after finalizing data collection.
  Differences between the two experimental groups regarding the frequencies of adverse events
Differences between the two experimental groups regarding the rates of revision due to aseptic loosening | 2 and 5 years after finalizing data collection.
  Differences between the two experimental groups regarding the rates of revision due to aseptic loosening

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Schilcher, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Universitetssjukhuset Linköping, Linköping, Region Östergotland, Sweden

IPD SHARING:
Plan to Share IPD: No